CLINICAL TRIAL: NCT05544071
Title: A Randomized, Sham-Controlled Trial Evaluating the Safety and Effectiveness of Precise Repetitive Transcranial Magnetic Stimulation (rTMS) Therapy Based on Neuroimaging in Depressed Adolescents With Anhedonia.
Brief Title: the Safety and Effectiveness of Precise rTMS Based on Neuroimaging in the Treatment of Adolescent Depression With Anhedoniadepression With Anhedonia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KY20222165-F-1
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Major Depressive Disorder; Repetitive Transcranial Magnetic Stimulation
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rTMS Active (Active Comparator): Blinded Active TMS coil. Active repetitive Transcranial Magnetic Stimulation (rTMS) and Sertraline (dosage form: pill, dosage: 50mg, frequency and duration: At the beginning of the treatment, the dose of 25mg/ was taken for 1-3 days and adjusted to 50mg/ days for 4-7 days. If there were no dose-limiting adverse events, the dose could be titrated to 100mg/ days in the second week. The dose could be flexibly adjusted within the range of 100~150mg/ days until a satisfactory clinical response was achieved. After that, the drug dose was kept unchanged as far as possible. Take it once a day, after a meal at a relatively fixed time in the morning.)
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)
- rTMS Sham (Sham Comparator): Blinded Sham TMS coil. Sham Transcranial Magnetic Stimulation (TMS) and Sertraline (dosage form: pill, dosage: 50mg, frequency and duration: At the beginning of the treatment, the dose of 25mg/ was taken for 1-3 days and adjusted to 50mg/ days for 4-7 days. If there were no dose-limiting adverse events, the dose could be titrated to 100mg/ days in the second week. The dose could be flexibly adjusted within the range of 100~150mg/ days until a satisfactory clinical response was achieved. After that, the drug dose was kept unchanged as far as possible. Take it once a day, after a meal at a relatively fixed time in the morning.)
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) — Compare active coil with sham coil.
  Other Names: TMS; Sertraline

SUMMARY:
This study evaluates a schedule of precise repetitive transcranial magnetic stimulation for depressive adolescent with anhedonia. In this randomized controlled trial, half of the participants will receive repetitive transcranial magnetic stimulation, and the other will receive sham stimulation.

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) is an established technology as therapy for treatment-resistant depression among adult. The approved method for treatment is 10Hz stimulation over the left dorsolateral prefrontal cortex (L-DLPFC). This methodology has been successful for many people with treatment-resistant depression. However, a large percentage of adolescents suffering from major depressive disorder (MDD) do not adequately benefit from currently available treatments. One of the limitations is concerns about the safety and efficacy of antidepressant. Recently, researchers have aggressively pursued better treatment strategy such as rTMS to improve adolescent depression with some preliminary success. This study intends to further explore the safety and efficacy of rTMS in the treatment for adolescent major depressive disorder with anhedonia. This study will also look at the change in neuroimaging biomarkers associated with this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 13 to 18 years of age.
* According to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Diagnosed with Major Depressive Disorder (MDD) and currently experiencing a Major Depressive Episode (MDE).
* Meet the threshold on the total HAMD17 score of >/=17 at both screening and baseline visits (Day -7 and Day 0).
* Meet the threshold on the total SHAPS score of >/=20 at both screening and baseline visits (Day -7 and Day 0).
* Not take any antidepressants for two or more weeks before screening.
* In good general health, as ascertained by medical history.
* After fully understanding the treatment of transcranial magnetic stimulation, willing to cooperate with the treatment actively and able to provide informed consent.

Exclusion Criteria:

* Current diagnosis of a Substance Use Disorder, with the exception of nicotine and caffeine dependence.
* Current diagnosis of mental disorders other than Dysthymic Disorder, Generalized Anxiety Disorder, Social Anxiety Disorder, Panic Disorder, Agoraphobia, or Specific Phobia (unless one of these is clinically unstable, and/or the focus of the participant's treatment for the past six months or more).
* History of schizophrenia or schizoaffective disorders, or any history of psychotic symptoms in the current or previous depressive episodes.
* Any other Mental Disorders, Personality Disorders, Intellectual Disability, which at screening is clinically predominant to their MDD.
* Has a clinically significant abnormality on the screening examination that might affect safety, study participation, or confound interpretation of study results.
* Any current or past history of any physical condition which in the investigator's opinion might put the subject at risk or interfere with study results interpretation.
* Participation in any clinical trial with an investigational drug or device within the past month or concurrent to study participation.
* History of electronic instrument or metal in the head or skull.
* History of epilepsy.
* History of cardiovascular disease or cardiac event.
* History of OCD.
* History of autism spectrum disorder.
* History of rTMS exposure.
* Other situations judged by the researchers to be unsuitable for the study.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 88 (Estimated)
Dates: Start 2023-02-12 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Percent Change in the Snaith-Hamilton Pleasure Scale (SHAPS)Score From Pre-treatment to 8-weeks | Pre-treatment and 8-weeks post treatment
  A 14 item self-assessment questionnaire used to measure the severity of anhedonia symptom in patients with mood disorders. Scale range - 14 to 56 with higher score indicative of greater anhedonia symptomology.

SECONDARY OUTCOMES:
Percent Change in the Hamilton Rating Scale for Depression (HAM-17) | Pre-treatment to 1 week and 15days, 4 weeks, 6 weeks and 8 weeks post-treatment
  A provider administered questionnaire used to assess remission and recovery from depression. Scale range - 0 to 52 with higher score indicative of greater depressive symptomology. Additional collection time points were prespecified; only those time points for which data were collected are reported.
Percent Change in the Montgomery Asberg Depression Rating Scale (MADRS) | Time Frame: Pre-treatment to 1 week and15days, 4 weeks, 6 weeks and 8 weeks post-treatment
  A diagnostic questionnaire used to measure the severity of depressive symptoms. Scale range - 0 to 60 with higher score indicative of greater depressive symptomology.
Percent Change in the Chinese version of Temporal Experience of Pleasure Scale(CV-TEPS) | Time Frame: Pre-treatment to 1 week and 15days, 4 weeks, 6 weeks and 8 weeks post-treatment
  A 20 item self-assessment questionnaire, eleven items used to measure anticipatory anhedonia, and nine items used to evaluate consummatory anhedonia. Scale range - 0 to 140 with lower score indicative of greater anhedonia symptomology.
Percent Change in the Chinese version of Beck Scale for Suicide Ideation（BSI-CV） | Time Frame: Pre-treatment to 1 week and 15days, 4 weeks, 6 weeks and 8 weeks post-treatment
  A 19 item questionnaire used to evaluate the severity of suicidal ideation. The scale includes two subscales of suicidal ideation (Current suicidal ideation, BSI-C) and suicidal ideation (Suicidal ideation at one's worst point, BSI-W) in the last week. Scale range - 0 to 38, the higher the score of the subscale, the higher the level of suicidal ideation in the last week or the most serious.
Percent Change in the Insomnia Severity Index Scale （ISI） | Time Frame: Pre-treatment to 1 week and 15days, 4 weeks, 6 weeks and 8 weeks post-treatment
  The questionnaire consists of seven items: the severity of insomnia symptoms, the satisfaction of sleep patterns, the effects of insomnia on daytime function, the effects of insomnia on subjects' quality of life, and the degree of worry or depression caused by insomnia. Scale range - 0 to 28 with higher score indicative of greater Insomnia symptomology.
Percent Change in the Clinical Global Impression (CGI) | Time Frame: Pre-treatment to 1 week and 15days, 4 weeks, 6 weeks and 8 weeks post-treatment
  The questionnaire used to evaluate the clinical efficacy, it includes three parts: severity of illness (SI), global improvement (GI) and effect index (EI). With higher score indicative of more serious disease and worse effect.
Percent Change in the Snaith-Hamilton Pleasure Scale (SHAPS) | Time Frame: Pre-treatment to 1 week and 15days, 4 weeks, 6 weeks and 8 weeks post-treatment
  A 14 item self-assessment questionnaire used to measure the severity of anhedonia symptom in patients with mood disorders. Scale range - 14 to 56 with higher score indicative of greater anhedonia symptomology.
Change From Baseline Functional Connectivity to 15-days Post-treatment | Time Frame: Pre-treatment, immediately post-treatment (on day 15)
  We will assess change in resting state fMRI functional connectivity of the nucleus accumbens to the Dorsolateral Prefrontal Cortex and within the reward-related circuits

OTHER OUTCOMES:
A digital tool named THINC-it® to help assess cognitive functioning | Time Frame: Pre-treatment to 1 week and 15days, 4 weeks, 6 weeks and 8 weeks post-treatment
  THINC-it® is a screening tool designed to measure cognition, is based on a combination of specific (traditional) neuropsychological tests assessing cognitive functioning, in conjunction with a patient-reported questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Zheng K, Chen L, Wang H; DIRECT consortium; Li B, Chen B. Beyond depression symptoms: the default mode network as a predictor of antidepressant response. Npj Ment Health Res. 2026 Jan 16;5(1):2. doi: 10.1038/s44184-025-00182-2. PMID 41545765
- [Derived] Lv R, Cai M, Tang N, Shi Y, Zhang Y, Liu N, Han T, Zhang Y, Wang H. Active versus sham DLPFC-NAc rTMS for depressed adolescents with anhedonia using resting-state functional magnetic resonance imaging (fMRI): a study protocol for a randomized placebo-controlled trial. Trials. 2024 Jan 13;25(1):44. doi: 10.1186/s13063-023-07814-y. PMID 38218932